CLINICAL TRIAL: NCT07154199
Title: Transcranial Ultrasound Stimulation for Cognitive Function Modulation in Patients With Post COVID-19 Brain Fog
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KS2022105-1
Record Dates: First submitted 2025-08-24; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: COVID-19; Brain Fog; Long COVID; Transcranial Ultrasound Stimulation
MeSH Terms: conditions — COVID-19; Mental Fatigue; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sham stimulation group (Sham Comparator): In the sham group, the transducer power was turned off, pre-recorded pulse repetition sounds were played to control for auditory confounds. The equipment appearance is consistent with the device. Single stimulation, 60 seconds.
  Interventions: Device: sham transcranial ultrasound stimulation
- real TUS group (Experimental): Ultrasound stimulation was delivered using TPO-203 and H-104MR_4AA-4CH transducer (Sonic Concepts, Woodinville, WA, USA). The target free-field spatial peak pulse-average intensity was maintained at 33.85 W/cm². The stimulation target is the right inferior Insula, according the results from observational study.
  Interventions: Device: real transcranial ultrasound stimulation

INTERVENTIONS:
Device: sham transcranial ultrasound stimulation — In the sham group, the transducer power was turned off, pre-recorded pulse repetition sounds were played to control for auditory confounds. The equipment appearance is consistent with the test device. Single stimulation, 60 seconds.
  Arms: sham stimulation group
Device: real transcranial ultrasound stimulation — Ultrasound stimulation was delivered using TPO-203 and H-104MR_4AA-4CH transducer (Sonic Concepts, Woodinville, WA, USA). In the real stimulation group, theta-burst TUS (Yaakub et al., 2024; Yaakub et al., 2023) was performed with the following parameters: pulse duration = 20 ms; pulse repetition interval = 200 ms; total duration = 80 s. The target free-field spatial peak pulse-average intensity was maintained at 33.85 W/cm². The stimulation target was defined as the overlapping region between the source localisation results and the right inferior insula in the Destrieux atlas
  Arms: real TUS group

SUMMARY:
This study aims to investigate whether a specific brain region mediates the cognitive deficit in long COVID brain fog, and whether targeted modulation of this region can improve cognition.

In observational study, the objective was to identify potential intervention targets for patients with long COVID brain fog. A total of 120 patients with long COVID were enrolled. Brain fog (BF) severity was quantified using the Brain Fog Assessment (BFA). Participants completed a continuous random-dot motion (cRDM) task during 128-channel electroencephalography (EEG) and underwent structural MRI and standardized neuropsychological testing.

In interventional study, 40 participants with persistent BF symptoms were enrolled for transcranial ultrasound stimulation (TUS). On Day 1, participants completed the BFA and provided demographic data, then performed the baseline cRDM task; 20 minutes later, structural MRI and baseline resting-state MRI were acquired. On Day 2, participants received 60 seconds of TUS (active or sham) according to randomized allocation. Twenty minutes post-stimulation, an 8-minute resting-state MRI scan was obtained, followed immediately by the follow-up cRDM task.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have a history of COVID-19 infection (positive test results for either polymerase chain reaction or rapid antigen test) and report persistent brain fog (BF) symptoms at least 4 weeks after recovering from acute COVID-19.

Exclusion Criteria:

* 1. Presence of any symptoms of cognitive impairment or other neurological symptoms prior to COVID-19 infection;
* 2. Structural MRI revealing significant intracranial lesions or structural abnormalities;
* 3. Development of severe neurological complications after COVID-19 infection, including delirium, cerebrovascular diseases, encephalitis, and epilepsy;
* 4. Other disorders that may cause cognitive impairment, including Dementia, Schizophrenia spectrum disorders, stroke, Alzheimer's disease, and Parkinson's disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
false alarm rate change | Day 1, Day 2
  false alarm rate change
accuracy change | Day 1, Day 2
  accuracy change

SECONDARY OUTCOMES:
false alarm rate | Day 1
  false alarm rate
accuracy | Day 1
  accuracy
cRDM modeling metrics | Day 1
  cRDM modeling metrics
Neural activation pattern of EEG | Day 1
  Neural activation pattern of EEG
Brain structure indicator of MRI | Day 1
  Brain structure indicator of MRI
resting-state functional connectivity change in MRI | Day 1, Day 2
  resting-state functional connectivity change in MRI

CONTACTS AND LOCATIONS:
Overall Officials: Yi Tang, MD., PhD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (2):
- China (2):
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Shandong Daizhuang Hospital, Jining, Shandong

IPD SHARING:
Plan to Share IPD: No